CLINICAL TRIAL: NCT02476721
Title: Characteristics of Patients With Missed Pulmonary Embolism in the ED: A Three Year Experience
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christoph Keil, Dr.med.univ., University Hospital, Basel, Switzerland
Other Study IDs: EKNZ 2014-183
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Missed Pulmonary Embolism at the Emergency Department
Keywords: pulmonary embolism; emergency department
MeSH Terms: conditions — Pulmonary Embolism; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: detection of pulmonary embolism

SUMMARY:
The clinical presentation of acute pulmonary embolism ranges from mild dyspnea and cough to shock or sustained hypotension but it also may even be asymptomatic and diagnosed by imaging procedures performed for other purposes. (1) Depending on the clinical presentation, the case fatality rate for acute pulmonary embolism ranges from 1% up to 60%. Due to the often non-specific presentation, especially in mild to moderate acute pulmonary embolism PE is often underdiagnosed. Chest pain and shortness of breath are the two most common symptoms associated with pulmonary embolism, together these symptoms are responsible for approximately 10 million emergency department visits in the United States of America (US) (2). The aim of this study was to determine the sensitivity and specificity of diagnosing pulmonary embolism (PE) at the emergency department (ED) of the University Hospital Basel and the investigators have therefore retrospectively analyzed all cases with excluded or proven PE in our institution in the last three years. Data sets from the institute of radiology, the institute of pathology and the ED are consistently available from January 2011 until the present day and were screened for pulmonary embolism in discharge reports. Data from the ED include all patients between January 2011 and December 2013 that presented to the ED and received either an ECG or any form of thoracic imaging. Particular attention was paid to patients with PE in the discharge report. The third set of data includes all patients with PE as cause of death or as a secondary diagnosis in the autopsy report. After comparing the three sets of data to each other the investigators tried to determine the sensitivity and specificity of PE diagnosis at the ED respectively the rate of missed diagnoses. A PE was seen as missed if it is detected 24h after the patient presented to the ED or if it was detected at another department after the patient was transferred from the ED.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older,
* presented to the ED between January 2011 and March 2014,
* who received an ECG or any form of thoracic imaging.

Exclusion Criteria:

* patients below 18 years of age, as well as patients referred to the ED with suspected PE by departments within UHBS, other hospitals, or other healthcare providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patientes presented to the ED in the specified timeframe who are at risk for pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 1251 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
in hospital mortality | 30 days

SECONDARY OUTCOMES:
initial ED diagnosis | 24 hours
characteristics of patients with missed PE | 30 days